CLINICAL TRIAL: NCT07292272
Title: Halt Aging in Survivors of Blood Cancers: the HALTAging-1 Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 606-25-FB
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin Lymphoma; Leukemia; Lymphoid Leukemia; Multiple Myeloma; Myeloid Leukemia; Monocytic Leukemia; Non-hodgkin Lymphoma; Other Hematologic Condition
MeSH Terms: conditions — Hodgkin Disease; Leukemia; Leukemia, Lymphoid; Multiple Myeloma; Leukemia, Myeloid; Leukemia, Monocytic, Acute; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm-Supervised (Experimental): intervention arm incorporating virtually supervised moderate-intensity aerobic exercise and behavioral intervention/coaching to improve adherence
  Interventions: Behavioral: Supervised Exercise and Coaching
- Enhanced Usual Care-Virtual Gym (Active Comparator): enhanced usual care arm, where survivors will get access to virtual gym membership only.
  Interventions: Behavioral: Virtual Gym Membership

INTERVENTIONS:
Behavioral: Supervised Exercise and Coaching — Intervention arm incorporating virtually supervised moderate-intensity aerobic exercise and behavioral intervention/coaching to improve adherence
  Arms: Intervention Arm-Supervised
Behavioral: Virtual Gym Membership — This arm will get access to a virtual gym membership only
  Arms: Enhanced Usual Care-Virtual Gym

SUMMARY:
Older survivors of blood cancer are at a high risk of accelerated biological aging, which increases their risk of developing multiple aging-related conditions. Whereas physical exercise can improve overall health, older cancer survivors do not meet the recommended physical activity, highlighting the need to develop behavioral interventions to increase adherence. Several other knowledge gaps exist to implement exercise interventions in older survivors of blood cancer; the dose and duration of exercise necessary to slow biological aging in older blood cancer survivors remain unknown. To bridge these gaps in knowledge, we have designed a Phase 2 randomized control trial to test the effects of behavioral and exercise interventions on various outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years
2. A history of hematological malignancy
3. Participants must be able to and willingly give informed consent

Exclusion Criteria:

1. Patients receiving intensive induction or consolidation chemotherapy. Maintenance chemotherapy, or lower-intensity chemotherapy for an indolent hematological malignancy is allowed.
2. Neurodegenerative disease (e.g. Alzheimer's dementia), stroke, or uncontrolled psychotic disorders (e.g. schizophrenia or bipolar disorder) in the past 3 months if those disorders are considered significant enough to impair participation in the study.
3. Illnesses such as clinical evidence of decompensated heart failure, unstable angina, or orthopedic or neuromuscular disorders that could limit safe participation in aerobic exercise.
4. Cardiopulmonary exercise test results that preclude safe exercise (e.g., life-threatening arrhythmia, balance difficulties, peak VO2 <10 ml/kg/min).
5. Estimated life expectancy of less than 6 months (that precludes assessment of study primary endpoint).
6. Participants who do not plan to follow up at the participating center.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-07-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who adhered to the exercise regimen at 6-months post enrollment. | 6 Months from start of program
  Adherence will be measured by those who completed 120 minutes or more of moderate exercise per week based on Polar Heart Rate data and Exercise Diaries.
Percentage of participants who adhered to the exercise regimen at 12-months post enrollment. | 12 Months from start of program.
  Adherence will be measured by those who completed 120 minutes or more of moderate exercise per week based on Polar Heart Rate data and Exercise Diaries.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No